CLINICAL TRIAL: NCT01901952
Title: Lifestyle Improvement Through Food and Exercise (LIFE) Study
Brief Title: Lifestyle Improvement Through Food and Exercise (LIFE)Study
Acronym: LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Cook County Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DK092271-01 (NIH); R01DK092271-01 (NIH)
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes
Keywords: Self management diabetes intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Active Comparator)
  Interventions: Behavioral: Standard of Care control group
- Intensive education and support (Experimental)
  Interventions: Behavioral: Intensive education and lifestyle support

INTERVENTIONS:
Behavioral: Intensive education and lifestyle support — Group classes for 12 months (weekly for 4 months, biweekly for 4 months, monthly for 4 months), weekly peer supporter telephone calls, and diabetes education newsletters every 2 months.
  Arms: Intensive education and support
Behavioral: Standard of Care control group — Participants receive 2 diabetes education classes taught by a Certified Diabetes Educator. They also receive diabetes education newsletters every 2 months.
  Arms: Standard of care

SUMMARY:
The primary aim of the LIFE study is to compare low-income African American diabetes patients in a lifestyle intervention group with those in a standard of care control group on change in glycemic control at 12-months. We hypothesize that, on average, participants in the intervention group will achieve greater glycemic control at 12-months relative to their baseline A1c, than those in the control group.

DETAILED DESCRIPTION:
This project is a randomized controlled trial to test an innovative lifestyle intervention to achieve sustained improvements in glycemic control among low-income African American diabetes patients. The LIFE (Lifestyle Improvement through Food and Exercise) program is a diabetes self-management program focused on diet and exercise, informed by anthropological research on models of food and health among low-income African-Americans. Pilot work demonstrated that the LIFE Program is effective in improving glycemic control among low-income African Americans at 6-months. The main goal of the current study is to determine whether the LIFE Program can achieve sustained improvements in glycemic control for 12 months. The trial will randomize low-income African American adults with diabetes to a control group, which receives standard diabetes education, or an intervention group, which receives the LIFE Program (28 group meetings with peer support telephone calls) followed by a 6-month maintenance phase (quarterly group sessions with monthly peer support phone calls). The primary aim of the proposed research is to compare low-income African American diabetes patients receiving the LIFE Program with those in a standard of care control group on change in glycemic control at 12 months. Our primary hypothesis is that patients in the intervention group will achieve a change in A1c from baseline that is less than patients in the control group. Secondary aims are to compare low-income African American diabetes patients receiving the LIFE Program with those in a standard of care control group on (a) change in glycemic control at 18 months; (b) change in physical activity and total energy intake at 12 months; (c) change in physical activity and total energy intake at 18 months; and (d) to obtain estimates needed for a subsequent trial, including weight, blood pressure, and diabetes-related hospitalizations. For secondary aims we hypothesize that a) the intervention group will achieve a mean 18-month change in A1C that is less than the change in the control group; b) at 12 months, a greater proportion of intervention patients will have achieved the activity goal of 150 minutes of moderate activity per week, and the intervention group will achieve a greater reduction from baseline in mean total energy intake than the control group; and c) at 18 months, a greater proportion of intervention patients will have achieved the activity goal of 150 minutes of moderate activity per week, and the intervention group will achieve a greater reduction from baseline in mean total energy intake than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus (T2DM) and HbA1c > 7%;
* Patients must identify themselves as African American;
* Patients must be patients of Cook County Hospital ambulatory clinics;
* Primary care physician gives clearance for patient to participate in study and engage in moderate level physical activity.

Exclusion Criteria:

* BMI<18.5;
* Patient not on diabetes medication and with a HbA1c reading less than 7%
* End-stage renal disease, stroke with paresis, congestive heart failure (NYHA class 2-4), or other major end-organ complication of diabetes;
* Comorbid conditions limiting probable life span to <4 years (e.g. cancer, AIDS) or indication of end-stage complications of diabetes (kidney dialysis, or transplant, blindness, or lower extremity amputation);
* Receiving treatment for a major psychiatric disorder (i.e. schizophrenia);
* Unable to give informed consent;
* Under the age of 18;
* Has no access to a telephone (Phone contact is a critical component of the intervention).
* Cannot walk 2 blocks without stopping and resting.
* Impaired cognitive function as determined by mini-mental test.
* Lives in the same household as an active LIFE participant.
* Presence of sickle cell trait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2012-03; Primary Completion 2015-11-25 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | change from baseline to 12 months
  Finger prick on Afinion machine

SECONDARY OUTCOMES:
Physical Activity | change from baseline to 12 months
  An accelerometer is worn by participants for seven days. International-Physical Activity Questionnaire is administered at baseline, 6 months, 1 year, and 18 months.
Total Energy Intake | change from baseline to 12 months
  24-hour dietary food recalls
Physical Measures | change from baseline to 12 months
  Measurements of weight, waist circumference, and blood pressure.
Medications | change from baseline to 12 months
  Participants bring all medications to the clinic visit and medication and dosage is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lynch, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Cook County Health Clinics, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lynch EB, Mack L, Avery E, Wang Y, Dawar R, Richardson D, Keim K, Ventrelle J, Appelhans BM, Tahsin B, Fogelfeld L. Randomized Trial of a Lifestyle Intervention for Urban Low-Income African Americans with Type 2 Diabetes. J Gen Intern Med. 2019 Jul;34(7):1174-1183. doi: 10.1007/s11606-019-04894-y. Epub 2019 Apr 8. PMID 30963440
- [Derived] Lynch EB, Liebman R, Ventrelle J, Keim K, Appelhans BM, Avery EF, Tahsin B, Li H, Shapera M, Fogelfeld L. Design of the Lifestyle Improvement through Food and Exercise (LIFE) study: a randomized controlled trial of self-management of type 2 diabetes among African American patients from safety net health centers. Contemp Clin Trials. 2014 Nov;39(2):246-55. doi: 10.1016/j.cct.2014.09.003. Epub 2014 Sep 22. PMID 25245954